CLINICAL TRIAL: NCT03756454
Title: A Prospective, Double-blind, Randomized, and Controlled Clinical Trial to Compare the Effectiveness of Intravenous Bezlotoxumab (10 mg/kg) Versus Placebo in Decreasing Morbidity and Mortality in Patients With Fulminant Clostridioides Difficile Requiring Surgical Intervention.
Brief Title: Comparing the Effectiveness of IV Bezlotoxumab Versus Placebo in Decreasing Morbidity and Mortality in Patients With Fulminant C. Diff Requiring Surgery.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with enrollment and inability to guarantee further study drug supply after current supply expired.
Sponsor: Michael E Villarreal, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Michael E Villarreal, MD, Clinical Instructor House Staff - General Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018H0348
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Clostridia Difficile Colitis; Clostridium; Sepsis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous; Sepsis | interventions — bezlotoxumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomization will be performed per best common practice guidelines with a computer generated randomization process and hospital investigational pharmacy blinding processes into both a therapeutic arm (Bezlotoxumab) and a placebo (normal saline) arm of the study. All current standards of care will continue to be administered in these patients, regardless of their respective study arm. To control for the antibiotics administered, the patients will need to be stratified according to the standard-of-care antibiotics and balanced in regards to this variable. Current standard of care therapy at our institution for fulminant C. difficile colitis includes Vancomycin (both oral and rectal, if needed) and intravenous Metronidazole. Fulminant C. difficile colitis is defined, per our guidelines, as proven infection with hypotension/ shock, ileus, or megacolon.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Upon conclusion of the surgical intervention, the Anesthesia or nursing team will administer the trial medication, Bezlotoxumab, or the placebo, normal saline. Dosing is planned to be ten milligrams per kilogram, which is standard dosing for therapeutic Bezlotoxumab approved for use by the U.S. Food and Drug Administration. This dose will be administered as a one-time single-infusion dose administered over the span of one hour. The placebo administration of normal saline will be at the same dosing with a single-infusion over one hour. The patient will receive standard of care post-operative management and the information obtained from standard-of-care lab draws will be assessed throughout their hospital stay. The patient will be seen and evaluated in clinic in the post-operative period at the one month follow-up and either in clinic or via telephone at their three month and six month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bezlotoxumab (Experimental): Patients receiving Bezlotoxumab post-operatively.
  Interventions: Biological: Bezlotoxumab
- Normal Saline (Placebo Comparator): Patients receiving normal saline as a placebo post-operatively.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Bezlotoxumab — Patients receiving Bezlotoxumab post-operatively.
  Arms: Bezlotoxumab
Other: Normal Saline — Placebo
  Arms: Normal Saline

SUMMARY:
A new medication, Bezlotoxumab, has been approved for treatment of recurrent Clostridium difficile diarrhea by the U.S. Food and Drug Administration. The way this new medication works, is by binding the toxin produced by C. difficile bacteria and preventing damage to the large bowel. The toxin, and not the bacteria, is responsible for the damage, resulting in the clinical symptoms seen in patients. Sometimes, the infection can make a patient severely ill with organ failure and death. If severe enough, the infection requires surgery to remove the large bowel and allow the patient a better chance at recovery. Even with surgery and removal of the bowel, patients can continue to be severely ill and have a very high rate of mortality. The toxin that injures the large bowel has been shown to obtain access to systemic circulation because of the injury to the bowel. At this time, the investigators continue antibiotics and supportive care to help patients recover post-operatively, as the investigators do not have other interventions in this critical population. Bezlotoxumab is known to bind this toxin and stop it from causing further injury in the bowel; it has the potential to bind the systemic toxin to prevent further damage throughout the body. This study is proposing that this new medication, Bezlotoxumab, can be added to the current standard of care for severe infection that requires surgery, and result in a decrease of the complications associated with this disease process. In this study, some patients will receive the medication after surgery; others will receive extra fluid. The investigators will not know who received which in order to decrease any bias in the results. All participants will receive similar post-operative care and be monitored closely. When enough patients are enrolled in the study, the results will be evaluated.

DETAILED DESCRIPTION:
Study Design This will be an interventional prospective, randomized, double-blinded controlled trial performed at a single center. Prospective data will be collected of all consenting patients with a diagnosis of either initial or recurrent fulminant C. difficile colitis requiring surgical intervention. The data to be collected includes standard-of-care blood draws; no extra lab draws are planned for this trial. In the event labs are not drawn, the investigators will plan to obtain serum creatinine, total bilirubin, and platelet counts to continue SOFA score evaluations while the patient is in the surgical ICU. Consent will be obtained either from the patient or their legally authorized representative. Inclusion criteria will be all patients over the age of eighteen with diagnosed fulminant C. difficile colitis requiring surgical colectomy with end ileostomy. Surgical intervention will be determined by the operating surgeon at the time of initial consult assessment and during the follow-up assessments while the patient is hospitalized. Patients may be excluded on the account they are pregnant, prisoners/ incarcerated, have a history of congestive heart failure, or have received IVIG within 30 days of randomization to exclusion criteria.

Randomization will be performed per best common practice guidelines with a computer-generated randomization process and hospital investigational pharmacy blinding processes into both a therapeutic arm (Bezlotoxumab) and a placebo (normal saline) arm of the study. All current standards of care will continue to be administered in these patients, regardless of their respective study arm. To control for the antibiotics administered, the patients will need to be stratified according to the standard-of-care antibiotics and balanced in regards to this variable. Current standard of care therapy at our institution for fulminant C. difficile colitis includes Vancomycin (both oral and rectal, if needed) and intravenous Metronidazole. Fulminant C. difficile colitis is defined, per our guidelines, as proven infection with hypotension/ shock, ileus, or megacolon.

Upon conclusion of the surgical intervention, the Anesthesia or nursing team will administer the trial medication, Bezlotoxumab, or the placebo, normal saline. Dosing is planned to be ten milligrams per kilogram, which is standard dosing for therapeutic Bezlotoxumab approved for use by the U.S. Food and Drug Administration. This dose will be administered as a one-time single-infusion dose administered over the span of one hour. The placebo administration of normal saline will be at the same dosing with a single-infusion over one hour. The patient will receive standard of care post-operative management and the information obtained from standard-of-care lab draws will be assessed throughout their hospital stay. The patient will be seen and evaluated in clinic during the post-operative period at the one-month follow-up and either in clinic or via telephone at their three-month and six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old, diagnosed C diff colitis requiring surgical intervention

Exclusion Criteria:

* CHF previously diagnosed, pregnancy, prisoners/ incarcerated, previous administration of IVIG within 30-days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Mortality | 30-days
  Monitor for 30-day mortality

SECONDARY OUTCOMES:
Heart Failure | 30-days
  Monitor for development of heart failure
Respiratory Failure | 30-days
  Monitor for development of respiratory failure
Renal Failure | 30-days
  Monitor for development of renal failure
Hepatic Failure | 30-days
  Monitor for development of hepatic failure

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No